CLINICAL TRIAL: NCT00031616
Title: A Phase I/II Study Of NB1011 Administered Intravenously Daily For 5 Days Every 4 Weeks In Fluoropyrimidine-Resistant Metastatic Or Relapsed Colorectal Cancers
Brief Title: NB1011 in Treating Patients With Metastatic or Recurrent Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NewBiotics (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069205; NB-1011-1001; NCI-V01-1689
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2004-04

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

INTERVENTIONS:
Drug: brivudine phosphoramidate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I/II trial to study the effectiveness of NB1011 in treating patients who have metastatic or recurrent colorectal cancer that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of NB1011 in patients with fluoropyrimidine-resistant metastatic or recurrent colorectal cancer.
* Determine the safety and toxic effects of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.
* Determine the efficacy of this drug in these patients.

OUTLINE: This is a phase I dose-escalation study followed by a phase II study.

* Phase I: Patients receive NB1011 IV over 1 hour on days 1-5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of NB1011 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Additional patients receive NB1011 at the MTD as in phase I. Patients are followed at day 30 and then for 5 months.

PROJECTED ACCRUAL: A maximum of 25 patients will be accrued for the phase I portion of this study. A total of 15-25 patients will be accrued for the phase II portion of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic or recurrent colorectal adenocarcinoma that has progressed during or within 6 months of fluoropyrimidine-based therapy
* Prior treatment with irinotecan with or without fluorouracil
* Evaluable or measurable disease

  * Uni-dimensionally measurable disease allowed provided CEA is at least 2 times the upper limit of normal
* No meningeal or CNS metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 1.5 mg/dL (regardless of liver metastases)
* AST and ALT less than 1.5 times upper limit of normal (ULN) (3 times ULN if liver metastases present)
* PT and INR normal
* PTT normal

Renal:

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance greater than 50 mL/min

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No known hypersensitivity to NB1011 or any excipient or vehicle in its formulation
* No active or uncontrolled serious bacterial, viral, fungal, or parasitic infection
* No prior or concurrent alcohol abuse or dependency
* No other malignancy within the past 2 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No concurrent medical or psychological condition that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* Recovered from prior anticancer chemotherapy
* No concurrent fluoropyrimidine-based or thymidylate synthase inhibitor agents

Endocrine therapy:

* Not specified

Radiotherapy:

* Recovered from prior anticancer radiotherapy
* No concurrent radiotherapy except palliative radiotherapy (to control a fracture or pain) provided index lesions are not involved

Surgery:

* Recovered from prior anticancer surgery

Other:

* At least 30 days since prior investigational agents
* No other concurrent anticancer therapy
* No concurrent disulfiram

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-12

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. Pegram, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (2):
- United States (2):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California